CLINICAL TRIAL: NCT01422512
Title: A Phase III Open Label, Uncontrolled, Multi Center Study to Evaluate Safety and Immunogenicity of a Surface, Antigen, Inactivated, Influenza Vaccine Produced in Mammalian Cell Culture, Formulation 2011/2012, When Administered to Adult and Elderly Subjects
Brief Title: Safety and Immunogenicity of One Dose of a Surface, Antigen, Inactivated, Influenza Vaccine Produced in Mammalian Cell Culture Administered to Adult and Elderly Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V58_25S; 2010-024613-31 (EudraCT Number)
Record Dates: First submitted 2011-08-23; First posted 2011-08-24 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Influenza
Keywords: seasonal influenza; vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cell culture derived TIV (Experimental): single dose of cell culture derived seasonal trivalent influenza vaccine (TIV)
  Interventions: Biological: seasonal influenza vaccine

INTERVENTIONS:
Biological: seasonal influenza vaccine — Subjects received one single IM dose of trivalent Surface, Antigen, Inactivated, Influenza Vaccine Produced in Mammalian Cell Culture during the vaccination visit, according to the study protocol (follow-up period: until day 22) .
  Other Names: Optaflu

SUMMARY:
This study will evaluate safety and immunogenicity of surface, antigen, inactivated, influenza vaccine produced in mammalian cell culture when administered to adult and elderly subject.

ELIGIBILITY:
Inclusion Criteria:

1. Males and female volunteers of 18 years of age or older, mentally competent, willing and able to give written informed consent prior to study entry
2. Individuals able to comply with all the study requirements
3. Individuals in good health as determined by the outcome of medical history, physical examination and clinical judgment of the investigator

Exclusion Criteria:

1. Individuals with behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the subject's ability to participate in the study
2. Individuals with any serious chronic or acute disease including but not limited to: Medically significant Cancer , Medically significant advanced congestive heart failure (ie. NYHA class III and IV),Chronic obstructive pulmonary disease (COPD); Autoimmune disease (including rheumatoid arthritis, except for Hashimoto's thyroiditis that has been clinically stable for ≥ 5 years);Diabetes mellitus type I/II ;Advanced arteriosclerotic disease ;History of underlying medical condition such as major congenital abnormalities requiring surgery, chronic treatment, or associated with developmental delay (e.g., Down's syndrome);Acute or progressive hepatic disease; Acute or progressive renal disease; Severe neurological or psychiatric disorder; Severe asthma
3. Individuals with history of any anaphylactic reaction and/or serious allergic reaction following a vaccination
4. Individuals with known or suspected impairment/alteration of immune function resulting, for example, from:

   receipt of immunosuppressive therapy (any parenteral or oral corticosteroid or cancer chemotherapy/radiotherapy) within the past 60 days and for the full length of the study; receipt of immunostimulants; receipt of parenteral immunoglobulin preparation, blood products and/or plasma derivates within the past 3 months and for the full length of the study; suspected or known HIV infection or HIV-related disease
5. Individuals with known or suspected history of drug or alcohol abuse
6. Individuals with a bleeding diathesis or conditions associated with prolonged bleeding time that in the investigator's opinion would interfere with the safety of the subject
7. Female who are pregnant or nursing (breastfeeding) mothers or females of childbearing potential not planning to use acceptable birth control measures, for the whole duration of the study
8. Individuals with history or any illness that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subjects due to participation in the study
9. Individuals who within the past 6 months have had any seasonal or pandemic laboratory confirmed influenza disease
10. Individuals who have received any seasonal or pandemic influenza vaccine;
11. Individuals with any acute or chronic infections requiring systemic antibiotic treatment or antiviral therapy within the last 7 days
12. Individuals who have experienced fever (i.e., axillary temperature ≥ 38°C) within the last 3 days of intended study vaccination
13. Individuals participating in another clinical trial
14. Individuals who have ever received blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation in the past 12 weeks and for the full length of the study
15. Individuals who are part of study personnel or close family members conducting this study
16. BMI > 35 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2011-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Antibody response as measured by hemagglutination inhibition (HI) assay | 22 days
  Antibody response to each influenza antigen as measured by hemagglutination inhibition (HI) at 21 days post-immunization in adult and elderly subjects in complinace with the requirements of the current EU recommendations for clinical trials related to yearly licensing of influenza vaccines

SECONDARY OUTCOMES:
Antibody response as measured by single radial hemolysis (SRH) assay | 22 days
  Antibody response to each influenza antigen as measured by single radial hemolysis (SRH) at 21 days post-immunization in adult and elderly subjects in complinace with the requirements of the current EU recommendations for clinical trials related to yearly licensing of influenza vaccines
Number of subjects with solicited local and systemic reactions | 7 days post vaccination
  To evaluate the safety of a single intramuscular (IM) injection of Optaflu in adult and elderly subjects in compliance with the requirements of the current EU recommendations for clinical trials related to yearly licensing of influenza vaccines (CPMP/BWP/214/96)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Reisinger, Principal Investigator — Universität Rostock / Medizinische Fakultät
Locations (1):
- Universität Rostock / Medizinische Fakultät, Rostock, Germany

REFERENCES:
- [Derived] Loebermann M, Voss U, Meyer S, Bosse D, Fritzsche C, Klammt S, Frimmel S, Riebold D, Reisinger EC. Clinical trial to evaluate the safety and immunogenicity of a trivalent surface antigen seasonal influenza vaccine produced in mammalian cell culture and administered to young and elderly adults with and without A(H1N1) pre-vaccination. PLoS One. 2013 Aug 16;8(8):e70866. doi: 10.1371/journal.pone.0070866. eCollection 2013. PMID 23976960